CLINICAL TRIAL: NCT05278351
Title: Tislelizumab Plus Cetuximab and Irinotecan Comparing the Third-line Standard-of-care Selected by Researchers in the Treatment of Ras Wild-type Recurrent Refractory Metastatic Colorectal Cancer: A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Tislelizumab Plus Cetuximab and Irinotecan vs Third-line Standard-of-care in Refractory mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEC2
Record Dates: First submitted 2022-03-08; First posted 2022-03-14 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Tislelizumab 200mg, D1, D15, intravenous drip, Q4W and Cetuximab 500mg/m2, D1, D15, intravenous drip, Q4W and Irinotecan 180mg/m2, D1, D15, intravenous drip, Q4W
  Interventions: Drug: Tislelizumab Combined With Cetuximab and Irinotecan
- B (Active Comparator): Fruquinitinib 5mg QD D1-21, oral, Q4W or Regorafenib 160mg QD D1-21 oral, Q4W or Trifluridine Tipiracil Tablets 35mg/m2 BID D1-D5, D8-D12 oral, Q4W
  Interventions: Drug: Third-line regimens

INTERVENTIONS:
Drug: Tislelizumab Combined With Cetuximab and Irinotecan — Tislelizumab (an anti-PD-1 monoclonal antibody) Cetuximab (monoclonal antibody against EGFR) Irinotecan
  Other Names: TEC
  Arms: A
Drug: Third-line regimens — Trifluridinetipiracil or Regorafenib or Fruquintinib
  Arms: B

SUMMARY:
This is a multicenter, randomized, controlled, phase II study to evaluate the efficacy and safety of tislelizumab combined with cetuximab and irinotecan（group A） compared to third-line regimens selected by researchers（group B） in the treatment of Ras wild-type recurrent and refractory metastatic colorectal cancer. This study will include Ras wild-type colorectal cancer that failed at least second-line treatment inthe past, including chemotherapy (oxaliplatin, irinotecan, fluorouracil) with or without targeted drugs (cetuximab, bevacizumab). 87 patients will be randomly assigned to group A and group B according to 2:1. The enrollment time is expected to be 12 months and the follow-up is expected to be 24 months.

ELIGIBILITY:
Inclusion Criteria：

* Age≥18years；
* The ECOG PS score was≤1;
* Ras wild-type colorectal cancer diagnosed by histology and/or cytology has metastasis or recurrence that cannot be cured by surgery;
* Have received at least second-line systemic anti-tumor treatments for mCRC and failed, in which chemotherapy drugs can include fluorouracil, oxaliplatin or irinotecan; with or without targeted drugs, such as cetuximab or bevacizumab;
* At least one measurable lesion defined according to RECIST version 1.1;
* Patients with fertility must be willing to take efficient contraceptive measures during the study period and ≥ 120 days after the last administration of drugs; female patients have negative urine or serum pregnancy test results ≤ 7 days before the first administration of the study drugs;
* Fully understand and voluntarily sign the informed consent form;
* Organ function is good ≤ 7 days before randomization, as shown in the following:

  a.Blood transfusion or growth factor support within 2 weeks before enrollment are not allowed to meet the enrollment criteria: i. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9 / L; ii.Platelet count≥ 75 × 10^9 / L; iii.Hemoglobin≥9g/dL or 90g / L or 5.6mmol/l; b. Serum total bilirubin ≤1.5 times the upper limit of normal value(ULN); c. Aspartate aminotransferase (AST) and alanine aminotransferase(ALT) ≤2.5 times ULN, or ALT and/or AST ≤5 times ULN in patients with liver metastasis; d. Serum creatinine ≤ 1.5 times the upper limit of normal value(ULN); e. Partial prothrombin time (APTT) or prothrombin time (PT) ≤1.5 times ULN; f. Albumin ≥30g / L;

Exclusion Criteria:

* Any previous histological or hematological ctDNA test showed mismatch repair gene deletion (dMMR), microsatellite instability (MSI-H), BRAF mutant patients;
* Previous immunotherapy, including anti-PD-1, anti-PD-L1, anti-CTLA-4 or any cellular immunotherapy;
* There is active leptomeningeal disease or brain metastasis that is not well controlled;
* History of active autoimmune diseases or autoimmune diseases that may recur. Note: Patients with the following diseases are not excluded and can be further screened:

  1. Well controlled type I diabetes mellitus
  2. Hypothyroidism (controlled by hormone replacement therapy only)
  3. Well controlled celiac disease
  4. Skin diseases that do not require systematic treatment (e.g. vitiligo, psoriasis, hair loss)
  5. Any other disease that is not expected to recur without external triggers
* Any active malignant tumor ≤ 5 years before the first administration of the study drug, except the specific cancer studied in this trial and any locally recurrent cancer that has received radical treatment (such as excised basal cell or squamous cell skin cancer, cervical or breast cancer in situ);
* Any case requiring systemic treatment with corticosteroids (prednisone or equivalent > 10 mg / day) or other immunosuppressive drugs ≤ 14 days before the first administration of the study drug. Note: patients who have currently or previously used any of the following steroid regimens are not excluded:

  1. Adrenal replacement steroids (prednisone or equivalent ≤ 10 mg / day)
  2. Inhaled corticosteroids with very low local, eye, intra-articular, intranasal or systemic absorption
  3. Short term (≤ 7 days) prophylactic use of corticosteroids (e.g. for the treatment of contrast medium allergy) or for the treatment of non autoimmune diseases (e.g. delayed type hypersensitivity caused by contact allergens)
* There was uncontrolled diabetes, or over 3 grade hypoalbuminemia or >1 grade potassium, sodium or calcium abnormalities within 14 days before the first drug administration,
* History of interstitial lung disease, non infectious pneumonia or uncontrolled diseases, including pulmonary fibrosis, acute lung disease, etc;
* Urine routine examination showed that urinary protein was ≥ + +, and 24-hour urinary protein was > 1.0 g;
* Severe chronic or active infections (including tuberculosis infection) requiring systemic antibacterial, antifungal or antiviral treatment within 14 days before the first administration of the study drug note: Patients with viral hepatitis are allowed to receive antiviral treatment;
* Active mental system diseases (schizophrenia, severe depressive disorder, bipolar disorder, etc.). Depression being treated with antidepressants is not an exclusion criterion;
* Known history of human immunodeficiency virus (HIV) infection;
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU / ml) or active HCV carriers with detectable HCV RNA. Note: carriers of inactive hepatitis B surface antigen (HBsAg) and patients with stable hepatitis B (HBV DNA < 500 IU / ml) can be included in the group;
* Any major surgery requiring general anesthesia ≤ 28 days before the first administration of the study drug;
* Previous heterologous stem cell transplantation or organ transplantation;
* Any of the following cardiovascular criteria

  1. Cardiogenic chest pain ≤ 28 days before the first administration of the study drug was defined as moderate pain limiting the movement of daily living instruments
  2. Symptomatic pulmonary embolism ≤ 28 days before the first administration of the study drug
  3. There was any history of acute myocardial infarction ≤ 6 months before the first administration of the study drug
  4. There was any history of heart failure with NYHA grade III or IV (6) ≤ 6 months before the first administration of the study drug
  5. There were any ventricular arrhythmia events with severity ≥ 2 ≤ 6 months before the first administration of the study drug
  6. There was any history of cerebrovascular accident ≤ 6 months before the first administration of the study drug
  7. Left ventricular ejection fraction (LVEF) ≤ lower normal limit (LLN) assessed by multi gated acquisition (MUGA) scan or echocardiography (echo). Follow up assessments must be performed in the same way as the baseline assessment
  8. Any syncope or seizure occurring ≤ 28 days before the first administration of the study drug
* Hypertension with poor control after multiple drug treatment (defined as systolic blood pressure > 140 mmHg and / or diastolic blood pressure > 90 mmHg);
* Hypersensitivity to any component of the study drug or control drug or to any component of the container;
* Bleeding, thrombotic disease or use of anticoagulants (such as warfarin) or similar drugs requiring therapeutic INR monitoring within 6 months before the first administration of the study drug;
* Chemotherapy, targeted therapy, immunotherapy (e.g. interleukin, interferon, thymosin, etc.), hormone therapy or any study therapy were performed within 14 days of the first administration of the study drug or within 5 half lives, whichever is shorter;
* Any Chinese herbal medicine or proprietary Chinese medicine with anticancer activity approved by China National Drug Administration within 14 days before the first administration of the study drug (regardless of cancer type);
* Toxicity from previous anticancer treatments did not improve to baseline or stable, except for AEs that were not considered as safety risks (e.g., hair loss, neuropathy and specific laboratory abnormalities);
* Live vaccine was administered ≤ 28 days before the first administration of the study drug.
* Potential disease conditions (including laboratory abnormalities), alcohol or drug abuse or dependence, which are not conducive to the administration of the study drug or affect the interpretation of the toxicity and AE of the study drug, or lead to insufficient or reduced compliance with the study;
* Participate in another clinical study at the same time, unless it is an observational (non intervention) clinical study or is in the follow-up period of intervention study;
* Inability to swallow capsules or diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, total gastrectomy or small bowel resection, weight loss surgery, inflammatory bowel disease or incomplete or complete intestinal obstruction;
* Uncontrollable pleural effusion, pericardial effusion or peritoneal effusion requiring frequent drainage or medical intervention within 7 days of the first administration of the study drug (clinically significant recurrence, additional intervention is required within 2 weeks after the intervention, excluding exfoliative cytology of the exudate);
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival time (PFS) | 24 months after the last subject participating in
  time from the start of medication to the initial progression of the disease

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months after the last subject participating in
  proportion of patients with complete and partial remission in the best efficacy
Disease control rate (DCR) | 24 months after the last subject participating in
  the best efficacy is the proportion of patients with complete remission, partial remission and stable disease
Overall survival (OS) | 36 months after the last subject participating in
  time from the start of medication to death

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes